CLINICAL TRIAL: NCT06388590
Title: Acupuncture for Chronic Pelvic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Moss (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Moss, Principal Investigator/MD, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MOMMC.2024.0029
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Pain; Acupuncture; Gynecology
Keywords: integrative medicine; acupuncture
MeSH Terms: conditions — Pelvic Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patient sample will be both control and treatment groups. Individuals will not be divided into distinct groups. Patients will serve as their own controls. Control patients will be participating in standard of care therapies including physical therapy, psychotherapy, behavioral health, typical primary care management, etc. as deemed appropriate by the primary care provider for 4 weeks prior to study intervention. The same patients will then be re-evaluated and will be offered Acupuncture with Dragon technique (see attachment Protocol for Needle Insertion) as a means of pain control once per week for 4 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Cohort: Control (Experimental): Patient sample will be both control and treatment groups. Individuals will not be divided into distinct groups. Patients will serve as their own controls. Control patients will be participating in standard of care therapies including physical therapy, psychotherapy, behavioral health, typical primary care management, etc. as deemed appropriate by the primary care provider for 4 weeks prior to study intervention. The same patients will then crossover and be re-evaluated and will be offered Acupuncture with Dragon technique (see attachment Protocol for Needle Insertion) as a means of pain control once per week for 4 weeks.
  Interventions: Other: Standard of Care
- Patient Cohort: Intervention (Experimental): Patient sample will be both control and treatment groups. Individuals will not be divided into distinct groups. Patients will serve as their own controls. Control patients will be participating in standard of care therapies including physical therapy, psychotherapy, behavioral health, typical primary care management, etc. as deemed appropriate by the primary care provider for 4 weeks prior to study intervention. The same patients will then crossover and be re-evaluated and will be offered Acupuncture with Dragon technique (see attachment Protocol for Needle Insertion) as a means of pain control once per week for 4 weeks.
  Interventions: Other: Dragons

INTERVENTIONS:
Other: Dragons — The Dragons Script will be read to the subjects by the provider administering treatment. Subjects will receive their Acupuncture treatment with Dragons protocol.
  Arms: Patient Cohort: Intervention
Other: Standard of Care — Standard of care therapies including physical therapy, psychotherapy, behavioral health, typical primary care management, etc. as deemed appropriate by the primary care provider for 4 weeks prior to study intervention.
  Arms: Patient Cohort: Control

SUMMARY:
The objective of this study is to determine if alternative pain management strategies, namely acupuncture, may help reduce intensity of female pelvic pain compared to other pain control modalities. This research study will focus specifically on the Dragon's protocol of acupuncture which will seek to alleviate chronic non-endometriosis pelvic pain for women both with and without a history of sexual assault.

This study may support evidence for an inexpensive alternative means of treatment for patients with or without traumatic sexual history and chronic pelvic pain.

DETAILED DESCRIPTION:
The objective of this study is to determine if alternative pain management strategies, namely acupuncture, may help reduce intensity of female pelvic pain compared to other pain control modalities. This research study will focus specifically on the Dragon's protocol of acupuncture which will seek to alleviate chronic non-endometriosis pelvic pain for women both with and without a history of sexual assault. The Dragons protocol consists of two parts, both completed at the same visit; external Dragons (needles are placed on the dorsal surface of the body) and internal Dragons (needles are placed on the ventral surface of the body). In Chinese Acupuncture theory, external dragons represent the traumatic events that happen in our life and the internal dragons represent dragons that live in the body and fight off the external dragons. It is used to treat post-traumatic stress. During external dragons the patient thinks about prior trauma (let the external dragons in) then during the second phase of treatment the internal dragons fight off the external dragons. From a western neurobiology perspective, clinical experience suggests that patients with post-traumatic stress have memories stored in the limbic system, that when triggered, activate the sympathetic nervous system. Dragons allows the brain to "reprocess" these memories so that triggers do not activate a sympathetic response in the patient. The mechanism is unknown, but the investigators theorize it may be due to vagal stimulation from the needles while the patient "relives" the traumatic event, thus experiencing the event in a parasympathetic state. This intervention will be compared to other treatment modalities such as pelvic floor physical therapy, non-steroidal anti-inflammatories, Osteopathic Manipulative Medicine, or any other usual means to achieve pain control offered by their providers.

The investigators will measure pre-procedure and post-procedure pain levels using the standard military Defense and Veterans Pain Rating Scale (DVPRS) in addition to a literature-based pelvic pain questionnaire, the Female Genitourinary Pain Index (GUPI). In addition to the pain index scales, patients with a history of sexual trauma will receive the PTSD Checklist for DSM-5 (PCL-5) which is a standardized measurement tool for assessing for PTSD. The provided acupuncture intervention, Dragon's, is classically used to treat both physical and emotional pain. Therefore, a sub-analysis will be performed to evaluate improvement in PTSD symptoms in those with a history of sexual assault and trauma.

The hypothesis of this study is that acupuncture with Dragon's will reduce chronic pelvic pain in females with and without a history of sexual trauma as it is designed to treat both physical and emotional pain. This is a relatively safe, effective, and non-invasive treatment strategy that could be offered as an alternative means of pain control when traditional modalities are ineffective.

Screening visit (30 minutes)

* Obtain and document signed Informed Consent document and HIPAA Authorization
* Verify subject eligibility based on inclusion/exclusion criteria via medical record review
* Record all medications the subject is taking
* Collect demographic information to include DoD ID, age, race, gender, military status (active duty, reserve, retired, separated or dependent), history of sexual assault prior to onset of pelvic pain, history of mental health diagnoses (e.g. anxiety, depression, PTSD), prior treatments used to treat pelvic pain

Patient sample will be both control and treatment groups. Individuals will not be divided into distinct groups. Patients will serve as their own controls. Control patients will be participating in standard of care therapies including physical therapy, psychotherapy, behavioral health, typical primary care management, etc. as deemed appropriate by the primary care provider for 4 weeks prior to study intervention. The same patients will then be re-evaluated and will be offered Acupuncture with Dragon technique (see attachment Protocol for Needle Insertion) as a means of pain control once per week for 4 weeks. Pain outcomes will be assessed with Defense and Veterans Pain Rating Scale (DVPRS) and Female Genitourinary Pain Index (GUPI). For subjects with a history of sexual trauma, a sub analysis will assess symptom change before and after treatment with PTSD Checklist for DSM-5 (PCL-5).

Visit 1 (week 0) (may be same day as screening visit) (20 minutes):

* Administer DVPRS including supplemental quality of life questions
* Administer GUPI
* Administer PCL-5 to subjects with a history of sexual assault

Visit 2 (week 4) (60 minutes) (In-Person):

* Subjects will report which treatments they have received since the screening visit
* Administer DVPRS including supplemental quality of life questions
* Administer GUPI
* Administer PCL-5 Monthly to subjects with a history of sexual assault
* The Dragons Script will be read to the subjects by the provider administering treatment
* Subjects will receive their initial Acupuncture treatment with Dragons

Visit 3 (week 5) (60 minutes) (In-Person):

* Administer DVPRS including supplemental quality of life questions
* Administer GUPI
* Administer PCL-5 Weekly to subjects with a history of sexual assault
* The Dragons Script will be read to the subjects by the provider administering treatment (visits 3-5 the subject can elect to read the script themselves).
* Subjects will receive their second Acupuncture treatment with Dragons

Visit 4 (week 6) (60 minutes) (In-Person):

* Administer DVPRS including supplemental quality of life questions
* Administer GUPI
* Administer PCL-5 Weekly to subjects with a history of sexual assault
* The Dragons Script will be read to the subjects by the provider administering treatment (visits 3-5 the subject can elect to read the script themselves).
* Subjects will receive their third Acupuncture treatment with Dragons

Visit 5 (week 7) (60 minutes) (In-Person):

* Administer DVPRS including supplemental quality of life questions
* Administer GUPI
* Administer PCL-5 Weekly to subjects with a history of sexual assault
* The Dragons Script will be read to the subjects by the provider administering treatment (visits 3-5 the subject can elect to read the script themselves).
* Subjects will receive their fourth Acupuncture treatment with Dragons

Visit 6 (week 11) (60 minutes) May be done virtually:

* Administer DVPRS including supplemental quality of life questions
* Administer GUPI
* Administer PCL-5 Monthly to subjects with a history of sexual assault

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Active Duty and DoD Female Beneficiaries (i.e. former military, spouse, dependent) aged 21-65 with chronic pelvic pain
* Have negative laparoscopic findings for endometriosis

Exclusion Criteria:

* Severe mental health disorders to include any disorder with psychotic features (e.g schizophrenia, bipolar, schizoaffective disorder)
* Pelvic pain as a result of severe physical trauma (excluding sexual assault) such as traumatic childbirth, pelvic fractures or any other trauma as determined by the PI or AI.
* Pregnancy

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Defense and Veterans Pain Rating Scale (DVPRS) | Visit 1 (Week 0)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | Visit 2 (Week 4)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | Visit 3 (Week 5)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | Visit 4 (Week 6)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | Visit 5 (Week 7)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | Visit 6 (Week 11)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Female Genitourinary Pain Index (GUPI) | Visit 1 (Week 0)
  GUPI is a validated instrument to assess the degree of symptoms in both men and women with genitourinary pain complaints. It has a range of 0 to 45 and has also demonstrated linear scale qualities allowing parametric methods to be used.
Female Genitourinary Pain Index (GUPI) | Visit 2 (Week 4)
  GUPI is a validated instrument to assess the degree of symptoms in both men and women with genitourinary pain complaints. It has a range of 0 to 45 and has also demonstrated linear scale qualities allowing parametric methods to be used.
Female Genitourinary Pain Index (GUPI) | Visit 3 (Week 5)
  GUPI is a validated instrument to assess the degree of symptoms in both men and women with genitourinary pain complaints. It has a range of 0 to 45 and has also demonstrated linear scale qualities allowing parametric methods to be used.
Female Genitourinary Pain Index (GUPI) | Visit 4 (Week 6)
  GUPI is a validated instrument to assess the degree of symptoms in both men and women with genitourinary pain complaints. It has a range of 0 to 45 and has also demonstrated linear scale qualities allowing parametric methods to be used.
Female Genitourinary Pain Index (GUPI) | Visit 5 (Week 7)
  GUPI is a validated instrument to assess the degree of symptoms in both men and women with genitourinary pain complaints. It has a range of 0 to 45 and has also demonstrated linear scale qualities allowing parametric methods to be used.
Female Genitourinary Pain Index (GUPI) | Visit 6 (Week 11)
  GUPI is a validated instrument to assess the degree of symptoms in both men and women with genitourinary pain complaints. It has a range of 0 to 45 and has also demonstrated linear scale qualities allowing parametric methods to be used.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Visit 1 (Week 0)
  Will be administered to subjects with history of sexual trauma.
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD Checklist for DSM-5 (PCL-5) | Visit 2 (Week 4)
  Will be administered to subjects with history of sexual trauma.
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD Checklist for DSM-5 (PCL-5) | Visit 3 (Week 5)
  Will be administered to subjects with history of sexual trauma.
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD Checklist for DSM-5 (PCL-5) | Visit 4 (Week 6)
  Will be administered to subjects with history of sexual trauma.
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD Checklist for DSM-5 (PCL-5) | Visit 5 (Week 7)
  Will be administered to subjects with history of sexual trauma.
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.
PTSD Checklist for DSM-5 (PCL-5) | Visit 6 (Week 11)
  Will be administered to subjects with history of sexual trauma.
  PCL-5 is a 20-item self-reporting measure of PTSD rating how the respondent has been bothered by PTSD symptoms over the past month using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Responses are summed to a total score with higher scores indicate greater PTSD symptom severity. A total symptom severity score (range 0 - 80) can be obtained by summing the scores for each of the 20 items. Research suggests that a PCL-5 cutoff score between 31-33 is indicative of probable PTSD. A 5 - 10 point change represents reliable change (i.e., change not due to chance) and a 10 - 20 point change represents clinically significant change.

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data

REFERENCES:
- [Background] Ahangari A. Prevalence of chronic pelvic pain among women: an updated review. Pain Physician. 2014 Mar-Apr;17(2):E141-7. PMID 24658485
- [Background] Lamvu G, Carrillo J, Ouyang C, Rapkin A. Chronic Pelvic Pain in Women: A Review. JAMA. 2021 Jun 15;325(23):2381-2391. doi: 10.1001/jama.2021.2631. PMID 34128995
- [Background] Li PS, Peng XM, Niu XX, Xu L, Hung Yu Ng E, Wang CC, Dai JF, Lu J, Liang RN. Efficacy of acupuncture for endometriosis-associated pain: a multicenter randomized single-blind placebo-controlled trial. Fertil Steril. 2023 May;119(5):815-823. doi: 10.1016/j.fertnstert.2023.01.034. Epub 2023 Jan 27. PMID 36716811
- [Background] Zhu X, Hamilton KD, McNicol ED. Acupuncture for pain in endometriosis. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD007864. doi: 10.1002/14651858.CD007864.pub2. PMID 21901713